CLINICAL TRIAL: NCT04203433
Title: A Pilot, Open-Label Study in Subjects With Mild-to-Moderate Plaque Psoriasis to Investigate the Dosing Feasibility, Safety, Tolerability, and Preliminary Efficacy of a Four-Week Multi-dose Regimen of DLX105-DMP Administered to a Target Lesion
Brief Title: A Study of DLX105-DMP in Subjects With Plaque Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DelArrivo, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DLX105-DMP-201
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DLX105-DMP Multi-Dose Twice Weekly (Experimental): 4 Weeks of 1mg DLX105-DMP applied to a target lesion twice weekly
  Interventions: Drug: DLX105-DMP
- DLX105-DMP Multi-Dose Once Weekly (Experimental): 4 Weeks of 1mg DLX105-DMP applied to a target lesion once weekly
  Interventions: Drug: DLX105-DMP

INTERVENTIONS:
Drug: DLX105-DMP — 1mg applied to target lesion

SUMMARY:
A Pilot, Open-Label Study in Subjects with Mild-to-Moderate Plaque Psoriasis to Investigate the Safety, Tolerability, and Preliminary Efficacy of a Four-Week Multidose Regimen of DLX105-DMP Administered to a Target Lesion

ELIGIBILITY:
Key Inclusion Criteria:

* Signed and dated informed consent.
* Subjects aged 18-75 years.
* Male subject, or if female, must be surgically sterile, post-menopausal, or using acceptable birth control.
* Stable chronic mild-to-moderate plaque psoriasis.

Key Exclusion Criteria:

* Non-plaque-type psoriasis only (e.g., pustular, erythrodermic and guttate psoriasis, palmar, or plantar) at Screening.
* Drug-induced psoriasis (i.e., new onset or exacerbation from beta-blockers, calcium channel inhibitors or lithium) within 3 months prior to Day 1.
* Ongoing use of psoriasis treatments or inadequate duration of washout prior to Day 1

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Local Tolerability Sensations | Up to 4 Weeks
  4-point likert scale: 0 = none, 1 = mild, 2 = moderate, or 3 = severe
Local Site Application Assessment | Up to 4 Weeks
  Investigator Assessment of Site Application Area using a 5-point scale: 0 = no visible reaction to 4 = severe erythema with induration/vesicles
Adverse Events | Day 1 through End of Study (Up to 4 Weeks after Last Dose)
  Treatment Emergent Adverse Events
Local Investigator Global Assessment (IGA) | Day 1 through End of Study (Up to 4 Weeks after Last Dose)
  Local Investigator Global Assessment of Target Lesion, using a 5-point scale: 0 = clear to 5 = severe
Local Psoriasis Area Severity Index Sum of Scores (Local PASI SOS) | Day 1 through End of Study (Up to 4 Weeks after Last Dose)
  Local Psoriasis Area Severity Index Total Score for the Target Lesion, total score of 0 to 12.

SECONDARY OUTCOMES:
Pharmacokinetic Parameters | Day 1, Day 15, and Day 25
  DLX105 concentrations in samples collected over time
Immunogenicity Testing | Up to 4 Weeks after Last Dose
  Presence of antidrug antibodies and drug neutralizing antibodies in samples collected over time

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - DelArrivo Investigational Site, Alpharetta, Georgia
  - DelArrivo Investigational Site, Philadelphia, Pennsylvania
  - DelArrivo Investigational Site, San Antonio, Texas
  - DelArrivo Investigational Site, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No
There is no current plan to make individual participant data available to other researchers; however, if study results are published, then de-identified IPD may be made available in connection with the publication.